CLINICAL TRIAL: NCT03565016
Title: Consequences of At-risk Alcohol Consumption in ICU Patients : the Impact OH Study.
Brief Title: Consequences of At-risk Alcohol Consumption in ICU Patients
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Impact OH
Record Dates: First submitted 2018-03-30; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Abuse; Alcoholism
Keywords: Alcohol use disorders; agitation; intensive care unit; restlessness; alcohol withdrawal syndrome; alcohol-dependence; heavy drinking
MeSH Terms: conditions — Alcoholism; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no interventional study — no interventional study

SUMMARY:
At-risk drinking is known to cause a high incidence of alcohol withdrawal syndrome which has a high impact on morbidity and mortality.

DETAILED DESCRIPTION:
Alcohol-use disorder has a significant impact on morbidity in surgical intensive care units and is known to cause alcohol withdrawal syndrome which mortality can reach 50% if left untreated. The aim of the study was to assess the impact of alcohol use disorder on one-year mortality and adverse ICU outcomes such as agitation in a Medical Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients aged 18 years old or more admitted in ICU

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 18 years old or more admitted in ICU non-at-risk drinkers or at-risk drinkers according to the National Institute of Alcohol Abuse and Alcoholism criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2013-11-25 (Actual); Study Completion 2013-11-25 (Actual)

PRIMARY OUTCOMES:
One-Year Mortality | The primary outcome measure was assessed at one year after ICU discharge
  Assessment of mortality at one year after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mickael Vour'ch, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France